CLINICAL TRIAL: NCT00464789
Title: An Open-Label, Single-Dose, Randomized, 3-Period, Crossover, Bioequivalence Study Between Bazedoxifene/Conjugated Estrogens (Premarin Current Process) And Bazedoxifene/Conjugated Estrogens (Premarin New Process) In Healthy Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene/Conjugated Estrogens Combinations In Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-1120
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Menopause
Keywords: Postmenopausal
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP); Tablets

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogens 20 mg/0.625 mg tablet

SUMMARY:
Bazedoxifene/Conjugated Estrogens (BZA/CE) is an investigational drug that is being developed for treatment of menopause. The purpose of this trial is to compare a new manufacturing process for making BZA/CE to the current process by assessing the way it is absorbed into the blood.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 35 to 70 years
* Body mass index (BMI) in the range of 18.0 to 35.0 kg/m2 and body weight greater than or equal to 50 kg
* Healthy as determined by the investigator on the basis of medical history, physical examination, breast and gynecologic examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Any clinically important active condition of gynecologic, cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* History or current evidence of thrombophlebitis, thromboembolic disorders, or any coagulopathies.
* History of any clinically important drug allergy to conjugated estrogens (CE) or selective estrogen receptor modulators (SERMs).

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
PK results

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer